CLINICAL TRIAL: NCT01551121
Title: Assessment of an Automated Telesurveillance System on the Incidence of Serious Falls in Nursing Homes
Acronym: TELEHPAD
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I11 004
Record Dates: First submitted 2012-03-01; First posted 2012-03-12 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2016-03

CONDITIONS: The Elderly of 75 Years and Living in Nursing Homes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- intervention group: Patient in the "intervention group" will have camera installed in their room. These cameras can either work in visible or infrared range. They are physically linked to a server that will store and analyze images in real-time. The server works 24h/24 and 7d/7 and will send an alert to the care personnel via their computers and personal pagers if it detects an anomaly. Anomaly could be falls, high risk behavior (patient standing up on its bed), abnormal length of stay in the bathroom, prolonged inertia. It will then allow them to intervene at the right time and the right place. Geriatrician can also review images in order to determine the cause of the incident and then act on each patient prevention and care strategy
  Interventions: Other: It will then allow them to intervene at the right time and the right place
- non-equipped group: Patient in the "non-equipped" group will have usual care
  Interventions: Other: It will then allow them to intervene at the right time and the right place

INTERVENTIONS:
Other: It will then allow them to intervene at the right time and the right place — The server works 24h/24 and 7d/7 and will send an alert to the care personnel via their computers and personal pagers if it detects an anomaly. Anomaly could be falls, high risk behavior (patient standing up on its bed), abnormal length of stay in the bathroom, prolonged inertia. It will then allow them to intervene at the right time and the right place. Geriatrician can also review images in order to determine the cause of the incident and then act on each patient prevention and care strategy.

SUMMARY:
3 Nursing homes in the Limousin region will be equipped with the automated telesurveillance system. Patient will be selected by general practitioner and randomized into two groups after informed consent. One group will have cameras installed and the other will not and will act as a comparison group. Patient will be assessed three times during the study, at inclusion, 6 months and 12 months. Each assessment is composed of a standard geriatric assessment, a fall questionnaire, an autonomy scale (SMAF scale) and a quality of life questionnaire (EQ5D). Every falls will be considered as adverse events and will therefore be listed along the study and characterized in types and number.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged more than 75 years old
* Patient living in Limoges or Gueret nursing home
* Patient informed consent and/or proxy consent
* Patient able to understand the study, respect its imperatives and able to do evaluations
* Patient able to stand up from the bed
* Patient covered by the French health insurance

Exclusion Criteria:

* Patient with a short term prognosis pathology
* In multiple bed rooms, if at least one patient does not agree with the trial

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: old subject
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The impact of the automated telesurveillance system on the risk ratio of falls | one year
  The impact of the automated telesurveillance system on the risk ratio of falls with serious outcomes between the two groups at one year

SECONDARY OUTCOMES:
The impact of the system on global risk of falling | 1 year
The impact of the system on autonomy loss | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thierry DANTOINE, MD, Study Director — University Hospital, Limoges; Michel PAILLER, MD, Principal Investigator — Gueret Hospital
Locations (1):
- Limoges University hospital, Limoges, France